CLINICAL TRIAL: NCT02718209
Title: The Development of an In-vitro System to Identify Gynecologic Cancer Cells During Surgical Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HYMC-84-15
Record Dates: First submitted 2016-03-21; First posted 2016-03-24 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Gynecological Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Frozen section (Experimental): Frozen sections taken from women operated on for possible gynecologic malignancies.
  Interventions: Device: Mid-Infrared Spectroscopy with ATR

INTERVENTIONS:
Device: Mid-Infrared Spectroscopy with ATR

SUMMARY:
The purpose of this study is to examine the efficacy of mid-infrared spectroscopy together with Attenuated Total Reflection (ATR), for the detection of gynecological malignancies in real time during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women with one or more tumors in reproductive system

Exclusion Criteria:

* Pregnant women
* Unable to give consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Gynecological Malignancies Identified in Real Time | One hour
  Results of Spectroscopy will be compared to frozen section/histopathology findings

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Bruchim, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No